CLINICAL TRIAL: NCT01867918
Title: A Randomized Study With Palliative Chemotherapy With or Without Local Treatment of Liver Metastases in Patients With Colo-rectal Cancer
Brief Title: LOTCOL Study: Local Treatment of Colo-rectal Liver Met
Acronym: LOTCOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insuffisient recruitment
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1392 REK South East C; 2012/1392 REK South East C
Record Dates: First submitted 2013-05-03; First posted 2013-06-04 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Radiofrequency Ablation; Microwaves; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cheomotherapy and local treatment (Experimental): Standard chemotherapy + local treatment
  Interventions: Procedure: Radiofrequency ablation, microwave, radiation therapy
- Cheomotherapy (Placebo Comparator): Standard chemotherapy
  Interventions: Drug: Standard Chemotherapy

INTERVENTIONS:
Procedure: Radiofrequency ablation, microwave, radiation therapy — Radiofrequency ablation Microwave ablation Radiation therapy
  Arms: Cheomotherapy and local treatment
Drug: Standard Chemotherapy
  Arms: Cheomotherapy

SUMMARY:
In this study the investigators will include colo-rectal cancer (CRC) patients starting last line of standard palliative chemotherapy. Eligible patients include patients with KRAS mutation starting line or KRAS wild type starting line treatment. Standard treatment today for these patients is chemotherapy only and median overall survival (OS) is about 10 months. The hypothesis is that local treatment in addition to systemic treatment will increase time to progression, progression free survival and overall survival compared to patients who receive systemic chemotherapy only. The investigators experience with local treatment of liver metastases in CRC patients is that side-effects of treatment in general are minor, although gastric bleeding have been observed after stereotactic body radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma of colon or rectum
* Ambulatory with an ECOG performance status 0-2
* At least 18 years of age
* Non-resectable liver metastases
* Progressive disease on or within 4 months after 1.line chemotherapy for KRAS mutant or after 2.line chemotherapy in KRAS wild type patients
* 1-4 liver metastases with largest diameter of up to 6 cm on CT-scan
* Up to 20 lesions in liver with no more than 4 lesions larger than 4 cm
* The patients will start 2./3. line chemotherapy (KRAS mutant/KRAS wt)
* Laboratory values as the following:

  * ANC ³ 1.5 x 109/L
  * Platelets ³ 100 x 109/L
  * Hb ³ 9g/dL
  * Creatinine £ 2x upper limit of normal
  * Bilirubin < 2.0x the upper limit of normal
  * ASAT and ALAT £ 5x the upper limit of normal
  * Albumin levels > 30 g/L
  * INR<1.3
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations

Exclusion Criteria:

* Previous treatment with 2. or 3. line chemotherapy (KRAS mutant/KRAS wt)
* History of prior metastatic disease the last 3 years
* History of CNS or bone metastases
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia
* Largest liver mets >6 cm, more than 4 liver lesions >4 cm
* Pulmonary mets>3 cm
* Lymph node mets >2.5 cm
* Chemotherapy/radiation therapy or major surgery within the last 4 weeks before start of treatment
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Overall survival from time of randomization | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway